CLINICAL TRIAL: NCT05669963
Title: Role of Oral Lactoferrin in Prevention of Recurnt Bacterial Vaginosis in Third Trimester of Pregnancy
Brief Title: Role of Oral Lactoferrin in Prevention of Recurnt Bacterial Vaginosis in Pregnancy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rania Samy Mohamed Ezzat, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB #9639/5-7-2022
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Bacterial Vaginosis | Vaginal | Microbiology
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Lactoferrin

STUDY DESIGN:
Intervention Model Description: Assuming the cure rate was 70.8% vs 33.3% in intervention vs placebo group. At 80% power and 95 % CI, the estimated sample will be 66 cases, 33 cases in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): study group receiving lactoferrin (2 capsules/day for 5 days followed by further 10 consecutive days at the dosage of 1 capsule/day) by oral intake.(pravotinR).
  During follow-up period, all women ingested 1 capsule of lactoferrin or placebo per day, for 10 consecutive days per month.
  Interventions: Drug: lactoferrin
- control group (Placebo Comparator): not recieving lactoferrin
  Interventions: Drug: lactoferrin

INTERVENTIONS:
Drug: lactoferrin — study grop receiving lactoferrin (2 capsules/day for 5 days followed by further 10 consecutive days at the dosage of 1 capsule/day) by oral intake.(pravotin).
  And another group not reciving lactoferrin.(control group) During follow-up period, all women ingested 1 capsule of lactoferrin or placebo per day, for 10 consecutive days per month.
  Other Names: PRAVOTIN

SUMMARY:
lactoferrin is believed to modulate immunity and help in prevention of recurrent bacterial vaginosis.In this study, the role of lactoferrin is assessed during third trimester of pregnancy.

DETAILED DESCRIPTION:
This study will be conducted at Zagazig University Hospitals, Obestetrics and Gynecology department, Zagazig University ,outpatient clinic .Assuming the cure rate was 70.8% vs 33.3% in intervention vs placebo group. At 80% power and 95 % CI, the estimated sample will be 66 cases, 33 cases in each group.

Among enrolled women those who have symptome of bacterial vaginosis will be treated with standard antibiotic therapy (metronidazole 500 mg twice daily for 7 days) and women who have history of recurrent bacterial vaginosis randomly assigned to one of two study arms: study grop receiving lactoferrin (2 capsules/day for 5 days followed by further 10 consecutive days at the dosage of 1 capsule/day) by oral intake.(pravotinR).

And another group not reciving lactoferrin.(control group) During follow-up period, all women ingested 1 capsule of lactoferrin or placebo per day, for 10 consecutive days per month.(study group) .

- All participating women attended 3 visits (from T0 to T2) at the gynaecologic centres at recruitment (T0), swap will be repeated after one month (T1) and two months (T2). In each clinical examination, 2 vaginal swabs (for vaginal culture and Nugent score) will be collected. During the first visit (baseline), patient medical history was recorded, informed consent was signed and women were allocated into the two study arms. - The evaluation of efficacy is based on clinical cure rate of BV symptoms (defined as absence of vaginal discharge or itching), microbiological cure rate (defined as remission and vaginal microbiota improvement by restoration of healthy Nugent score with range 0-3), and overall cure rate (absence of symptoms and Nugent score <7). In addition, recurrence rate was calculated for both groups as percentage of women presenting with symptoms and Nugent score more than 3 during the follow-up period. Safety is assessed by recording all side effects (i.e. adverse events, serious adverse events, and suspected unexpected serious adverse reactions). An adverse event is considered severe if it was fatal, life threatening, required hospitalisation, or led to permanent injury.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women of age group 20-37 years.
2. Primigravida.
3. 28-40 week gestation.
4. History of receurent bacterial vaginosis .

Exclusion Criteria:

1. Multiple gestations.
2. Multiparity.
3. Medical disorders as:

   * Diabetes mellitus.
   * Chronic hypertension.
   * Endocrinal diseases.
   * Autoimmune diseases.
   * Renal diseases.
   * Blood diseases.
4. Allergy to lactoferrin .

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
clinical cure rate of bacterial vaginosis symptoms | 3 months
  clinical cure rate of bacterial vaginosis symptoms (defined as absence of vaginal discharge or itching)
microbiological cure rate of bacterial vaginosis | 3 months
  defined as remission and vaginal microbiota improvement by restoration of healthy Nugent score with range 0-3), and overall cure rate (absence of symptoms and Nugent score <7)
recurrence rate of bacterial vaginosis | 3 months
  recurrence of bacterial vaginosis symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rania Samy Ezzat, MD, Study Director — Lecturer of obstetrics and Gynecology, Faculty of Medicine, Zagazig University; Amal Mohamed Alanwar, MD, Study Chair — Professor of obstetrics and Gynecology, Faculty of Medicine, Zagazig University; Safaa Abdelsalam Ibrahim, MD, Study Director — Professor of obstetrics and Gynecology, Faculty of Medicine, Zagazig University; Marian Asaad Gerges, MD, Study Director — Assistant Professor of Microbiology and Immunology Faculty of Medicine Zagazig University; Khoulh Al Mahdi Anbeeh Al Barhami, MBBCH, Principal Investigator — Master's degree candidate
Locations (1):
- Rania Samy ezzat, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No